CLINICAL TRIAL: NCT01160458
Title: Phase II Study of IMC-A12 in Patients With Mesothelioma Who Have Been Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raffit Hassan, M.D., Dr. Raffit Hassan, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100146; 10-C-0146
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Results first posted 2013-05-14 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Pleural Mesothelioma; Peritoneal Mesothelioma
Keywords: Monoclonal Antibody; Pleural Mesothelioma; Peritoneal Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMC-A12 Monotherapy in Patients (Experimental): 20 mg/kg intravenous over 60 minutes or not to exceed 25 mg/minute once every 3 weeks (+ or -1 day cycle 3 and beyond)
  Interventions: Drug: IMC-A12

INTERVENTIONS:
Drug: IMC-A12 — 20 mg/kg intravenous over 60 minutes or not to exceed 25 mg/minute once every 3 weeks (+ or -1 day cycle 3 and beyond)
  Other Names: A12 Cixutumumab

SUMMARY:
Background:

Background:

- IMC-A12, a new cancer treatment that has not yet been approved by the U.S. Food and Drug Administration, is an antibody that is designed to block the effects of a protein called Type I Insulin-Like Growth Factor (IGF-1R). IMC-A12 blocks the receptors in cells that respond to IGF-1R, which are thought to play an important role in helping cancer cells to grow and divide. Researchers are interested in determining whether IMC-A12 is an effective treatment for individuals who have mesothelioma that has not responded to standard chemotherapy.

Objectives:

- To evaluate the safety and effectiveness of IMC-A12 treatment in individuals with mesothelioma who have previously had chemotherapy.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with mesothelioma that has not responded to chemotherapy.

Design:

* Eligible participants will be screened with a full physical examination and medical history, blood and urine samples, and imaging studies.
* Participants will receive IMC-A12 once every 3 weeks (21-day cycle), and will be evaluated before the start of each new cycle with blood tests and imaging studies if needed.
* Treatment cycles will continue for as long as needed, unless severe side effects develop or the disease progresses.

DETAILED DESCRIPTION:
Background:

Platinum-based chemotherapy is the standard of care for advanced unresectable malignant mesothelioma. New options for treatment are necessary in patients with advanced disease that have progressed on platinum-based therapy. The insulin-like growth factor (IGF) pathway is being studies in various malignancies including mesothelioma. IMC-A12 is an anti-IGF-1R monoclonal antibody that has shown activity in patients with various malignancies.

Objectives:

Primary Objective:

- To determine the clinical response rate (partial response (PR)+complete response (CR)) to IMC-A12 monotherapy in patients with advanced mesothelioma.

Secondary Objectives:

* To determine response duration, progression free survival (PFS) and overall survival (OS).
* To assess safety of IMC-A12 in patients with mesothelioma

Exploratory Objectives:

* To evaluate tumor IGF-1R expression and correlation with response
* To correlate response to therapy with changes in fludeoxyglucose 18F-positron emission tomography (FDG-PET) imaging.
* To monitor serum mesothelin and cancer antigen 125 or carbohydrate antigen 125 (CA-125) levels prior to and during therapy.

Eligibility:

* Patients with histologically confirmed malignant pleural or peritoneal mesothelioma who have previously been treated on at least one platinum-containing chemotherapy regimen with progressive disease documented prior to study entry, or have refused cytotoxic chemotherapy.
* Measurable disease by modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria for pleural mesothelioma or by RECIST criteria for peritoneal mesothelioma.
* Adequate renal, hepatic and hematopoietic function.
* No major surgery, radiotherapy, chemotherapy or biologic therapy within 28 days of IMC-A12 therapy

Design:

* Patients will receive IMC-A12 at a dose of 20 mg/kg intravenously once every three weeks.
* Treatment with IMC-A12 alone will continue until disease progression.
* Toxicity will be assessed every cycle by the Cancer Therapy Evaluation Program (CTEP) Version 4.0 of Common Terminology Criteria for Adverse Events (CTCAE).
* Tumor response assessments will be performed every 2 cycles.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Subjects must have histologically confirmed pleural or peritoneal mesothelioma not amenable to potentially curative surgical resection. The diagnosis will be confirmed by the pathology department / Center for Cancer Research (CCR) / National Cancer Institute (NCI).
2. Patients must have had at least one prior platinum-containing chemotherapy regimen. There is no limit to the number of prior chemotherapy regimens received.
3. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan.
4. Patients must not have had major surgery, radiation therapy, chemotherapy, biologic therapy (including any investigational agents), or hormonal therapy (other than replacement), within 4 weeks prior to entering the study and must have evidence of stable or progressive disease to be eligible.
5. Age greater than or equal to 18 years. Since mesothelioma is extremely rare in children they are excluded from this study.
6. Life expectancy of greater than 3 months.
7. Performance status Eastern Cooperative Oncology Group (ECOG) less than or equal to 2.
8. Patients must have adequate organ and marrow function (as defined below).

   * leukocytes greater than or equal to 3,000/mm^3
   * absolute neutrophil count greater than or equal to 1,500/mm^3
   * hemoglobin greater than or equal to 9 g/dL
   * platelets greater than or equal to 100,000/ mm^3
   * total bilirubin less than or equal to 1.5 times institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase(SGPT) less than or equal to 3 times institutional ULN

     (5 times if liver function test (LFT) elevations due to liver metastases)
   * creatinine less than or equal to 1.5 times institutional ULN

   OR

   - creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine

   levels above institutional normal

   Patients may be transfused to obtain a hemoglobin of greater than or equal to 9 g/Dl.
9. The patient must have fasting serum glucose < 160 mg/dL
10. The effects of IMC-A12 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) for the duration of study therapy and for 3 months after the last dose of IMC-A12. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. While hormonal methods of birth control are effective, we ask that female patients who are participating in the study cease hormonal forms of birth control, as these methods of birth control (birth control pills, injections, or implants) may affect the study drug. Patients must be off hormonal forms of birth control for at least 4 weeks prior to initiating the study.
11. Ability to comply with intravenous administration schedule, and the ability to understand and the willingness to sign a written informed consent document.

Inclusion of Women and Minorities

Both men and women and members of all races and ethnic groups are eligible for this trial. Every effort will be made to recruit women and minorities in this study.

EXCLUSION CRITERIA:

1. Patients with symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients who have had treatment for their brain metastases and whose brain metastatic disease status has remained stable for at least 3 months without steroids may be enrolled at the discretion of the principal investigator.
2. Patients with poorly controlled diabetes mellitus. Patients with a history of diabetes mellitus are allowed to participate, provided their blood glucose is below 160 mg/dL when fasting and if they are on a stable dietary or therapeutic regimen for this condition with their HbA1C of less than 7%.
3. Uncontrolled medical illness including, but not limited to, ongoing or uncontrolled, symptomatic congestive heart failure (American Heart Association (AHA) Class II or worse), uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Human immunodeficiency virus (HIV) positive patients with poorly controlled viral loads (viral load > 50 copies HIV/ml), and/or acquired immune deficiency syndrome (AIDS)-defining illnesses will be excluded due to the possibility that IMC-A12 may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events with respect to IMC-A12. HIV positive patients with mesothelioma not meeting the above criteria can be considered for inclusion in the study.
5. Patients may not be receiving any other investigational agents.
6. History of another invasive malignancy in the last five years. Adequately treated non-invasive, non-melanoma skin cancers as well as in situ carcinoma of the cervix will be allowed.
7. Prior treatment with drugs of the IGF-1R inhibitor class.
8. Patients with tumor amenable to potentially curative therapy as assessed by the investigator. In patients with peritoneal mesothelioma who have had no prior surgery, a surgical consultation will be obtained to see if the patient is a candidate for debulking surgery.
9. Pregnant women are excluded from this study because IMC-A12 is a monoclonal antibody to IGF-1R with the potential for teratogenic or abortifacient effects. Immunoglobulin G (IgG) antibody may also potentially be secreted in milk and therefore breastfeeding women should be excluded. Because of the potential of teratogenic or abortifacient effects women of childbearing potential and men must agree to use adequate contraception (barrier methods) before, during the study and for a period of 3 months after the last dose of the investigational agent.
10. Patients must not be on hormonal forms of birth control or hormone replacement therapy, as this may affect the study drug. Patients must be off hormonal forms of birth control or hormone replacement therapy for at least 4 weeks prior to initiating the study.
11. History of allergic reactions attributed to compounds of similar chemical or biologic composition to IMC-A12.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06-02 (Actual); Primary Completion 2016-08-13 (Actual); Study Completion 2017-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bridda A, Padoan I, Mencarelli R, Frego M. Peritoneal mesothelioma: a review. MedGenMed. 2007 May 10;9(2):32. PMID 17955087
- [Background] Vogelzang NJ, Rusthoven JJ, Symanowski J, Denham C, Kaukel E, Ruffie P, Gatzemeier U, Boyer M, Emri S, Manegold C, Niyikiza C, Paoletti P. Phase III study of pemetrexed in combination with cisplatin versus cisplatin alone in patients with malignant pleural mesothelioma. J Clin Oncol. 2003 Jul 15;21(14):2636-44. doi: 10.1200/JCO.2003.11.136. PMID 12860938
- [Background] O'Byrne KJ, Edwards JG, Waller DA. Clinico-pathological and biological prognostic factors in pleural malignant mesothelioma. Lung Cancer. 2004 Aug;45 Suppl 1:S45-8. doi: 10.1016/j.lungcan.2004.04.025. PMID 15261433
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0146.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMC-A12 Monotherapy in Patients
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IMC-A12 Monotherapy in Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.28 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate (PR+CR)
Description: Clinical response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is complete disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | IMC-A12 Monotherapy in Patients
Number analyzed (Participants) | 20
Participants
  Complete Response | 0
  Partial Response | 0

2. Secondary Outcome: Safety of IMC-A12 in Patients With Mesothelioma
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | IMC-A12 Monotherapy in Patients
Number analyzed (Participants) | 20
Participants | 20

3. Secondary Outcome: Duration of Overall Response
Description: Duration of Overall Response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Complete response is complete disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease is at least a 20% increase in the sum of the longest diameter of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 36 months
Population: No participants had a complete response or partial response.
Arm/Group | IMC-A12 Monotherapy in Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival is defined as the time interval from the start of treatment to documented evidence of disease progression. Progressive disease is at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study longest diameter (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: To study completion, an average of 3 years
Population: One participant withdrew from the study and was excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-A12 Monotherapy in Patients
Number analyzed (Participants) | 19
months | 1.8 [1.4 to 5.5]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is the time interval from the start of treatment to the date of death.
Time Frame: To study completion, an average of 3 years
Population: One participant withdrew from the study and was excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | IMC-A12 Monotherapy in Patients
Number analyzed (Participants) | 19
Months | 5.5 [2.1 to 12.2]

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 36 months.
Arm/Group | IMC-A12 Monotherapy in Patients
All-Cause Mortality (participants affected / at risk) | 16/20
Serious Adverse Events (participants affected / at risk) | 19/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 Monotherapy in Patients (N=20)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Alkaline phosphatase increased (Investigations) | 2 (3)
Allergic rhinitis (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Atrial flutter (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Confusion (Psychiatric disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (4)
Death NOS (General disorders) | 16 (16)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Dental caries (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 10 (11)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hypotension (Vascular disorders) | 3 (4)
Infections and infestations - Other, thrush (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, mailgnant and unspecified (incl cysts and polyps)-Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 Monotherapy in Patients (N=20)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (6)
Bloating (Gastrointestinal disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Investigations) | 5 (20)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 8 (8)
Fever (General disorders) | 2 (2)
Floaters (Eye disorders) | 4 (5)
Headache (Nervous system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (30)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (9)
Hyponatremia (Metabolism and nutrition disorders) | 8 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Oral pain (Gastrointestinal disorders) | 1 (2)
Platelet count decreased (Investigations) | 6 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sore throat (Gastrointestinal disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (6)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 12 (14)
Dizziness (Nervous system disorders) | 5 (5)
Dysphasia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT01160458/Prot_ICF_000.pdf